CLINICAL TRIAL: NCT03055689
Title: Nurse-led Educational Telephone Intervention for Bowel Preparation for Repeat Colonoscopy After Preparation Failure (RepeatPrep Study)
Brief Title: Bowel Preparation for Repeat Colonoscopy After Preparation Failure (RepeatPrep Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Hospital Universitario de Canarias (Other)
Responsible Party: Principal Investigator, Marco Antonio Alvarez Gonzalez, Gastroenterologist deputy doctor, MD, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REPEATPREP
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Bowel Preparation for Colonoscopy
Keywords: Colonoscopy; Educational intervention
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational telephone intervention (Experimental): This group will receive a nurse-led educational telephone intervention for bowel preparation 24-48 before the colonoscopy
  Interventions: Behavioral: Educational telephone intervention
- Standard education for colonoscopy (Active Comparator): The control group will receive standard education for bowel preparation at the time of colonoscopy scheduling
  Interventions: Behavioral: Standard education for colonoscopy

INTERVENTIONS:
Behavioral: Educational telephone intervention — Subjects will receive a nurse-led educational telephone intervention for bowel preparation 24-48 hours before the colonoscopy
  Arms: Educational telephone intervention
Behavioral: Standard education for colonoscopy — Standard education for bowel preparation at the time of colonoscopy scheduling
  Arms: Standard education for colonoscopy

SUMMARY:
This trial will evaluate the efficacy in colon cleansing of a nurse-led educational telephone intervention 24-48 hours before a colonoscopy, in selected participants with a previous inadequate bowel preparation.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with a colonoscopy with inadequate bowel preparation, for any indication and where the endoscopist considers that the colonoscopy should be repeated to optimize the visualization with a better bowel preparation. Participants must have been properly informed and they have to sign the inform consent.

Exclusion Criteria:

* Hospitalized patients
* Unwillingness to participate in the study
* Inability to follow instructions: cognitive impairment or language barrier
* Inability to use a telephone or not owning a telephone
* Active inflammatory bowel disease
* Severe renal impairment
* Pregnancy of breast feeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 657 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-25 (Actual)

PRIMARY OUTCOMES:
Adequate bowel cleansing for colonoscopy | At the moment of colonoscopy
  The efficacy of bowel preparation will be rated by blinded endoscopists using the Boston Bowel Preparation Scale (BBPS). Adequate bowel cleansing will be defined as a BBPS of 2 or more points in every segment of the colon and inadequate bowel cleansing will be defined by at least one of the colon segments with less than 2 points.

SECONDARY OUTCOMES:
Overall adenoma detection rate, as defined by the ratio of patients with at least one adenoma in the overall colon | At the moment of colonoscopy
  The ratio of patients with at least one adenoma in the overall colon
Adenoma detection rate in the right colon | At the moment of colonoscopy
  Ratio of patients with at least one adenoma in the right colon (proximal to the splenic flexure)
Overall serrated lesion detection rate | At the moment of colonoscopy
  Ratio of patients with at least one serrated lesion in the overall colon
Serrated lesion detection rate in the right colon | At the moment of colonoscopy
  Ratio of patients with at least one serrated lesion in the right colon (proximal to the splenic flexure)
Complete colonoscopy rate | At the moment of colonoscopy
  Ratio of successful complete colonoscopies (cecal intubation or in case of previous surgery, ileocolic anastomosis)
Boston Bowel Preparation Scale | At the moment of colonoscopy
  Application of the Boston Bowel Preparation Scale to evaluate colonoscopy bowel cleansing
Barcelona Bowel Preparation Scale | At the momento of colonoscopy
  Application of the Barcelona Bowel Preparation Scale to evaluate colonoscopy bowel cleansing

CONTACTS AND LOCATIONS:
Locations (14):
- Spain (14):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Althaia Hospital de Manresa, Manresa, Barcelona
  - Consorci Sanitari Terrassa, Terrassa, Barcelona
  - Hospital de Viladecans, Viladecans, Barcelona
  - Hospital Santos Reyes, Aranda de Duero, Burgos
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - Hospital Universtiario de Móstoles, Móstoles, Madrid
  - Hospital Del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital 12 de Octubre, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Santa Bárbara, Soria
  - Hospital Rio Hortega, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alvarez-Gonzalez MA, Flores-Le Roux JA, Seoane A, Pedro-Botet J, Carot L, Fernandez-Clotet A, Raga A, Pantaleon MA, Barranco L, Bory F, Lorenzo-Zuniga V. Efficacy of a multifactorial strategy for bowel preparation in diabetic patients undergoing colonoscopy: a randomized trial. Endoscopy. 2016 Nov;48(11):1003-1009. doi: 10.1055/s-0042-111320. Epub 2016 Aug 4. PMID 27490086
- [Result] Ness RM, Manam R, Hoen H, Chalasani N. Predictors of inadequate bowel preparation for colonoscopy. Am J Gastroenterol. 2001 Jun;96(6):1797-802. doi: 10.1111/j.1572-0241.2001.03874.x. PMID 11419832
- [Result] Ibanez M, Parra-Blanco A, Zaballa P, Jimenez A, Fernandez-Velazquez R, Fernandez-Sordo JO, Gonzalez-Bernardo O, Rodrigo L. Usefulness of an intensive bowel cleansing strategy for repeat colonoscopy after preparation failure. Dis Colon Rectum. 2011 Dec;54(12):1578-84. doi: 10.1097/DCR.0b013e31823434c8. PMID 22067188
- [Result] Liu X, Luo H, Zhang L, Leung FW, Liu Z, Wang X, Huang R, Hui N, Wu K, Fan D, Pan Y, Guo X. Telephone-based re-education on the day before colonoscopy improves the quality of bowel preparation and the polyp detection rate: a prospective, colonoscopist-blinded, randomised, controlled study. Gut. 2014 Jan;63(1):125-30. doi: 10.1136/gutjnl-2012-304292. Epub 2013 Mar 16. PMID 23503044